CLINICAL TRIAL: NCT02464683
Title: Effect of Vitamin D as Adjunctive Therapy in Patients With Pulmonary Evolution Tuberculosis in the National Institute of Respiratory Diseases
Brief Title: Effect of Vitamin D as Adjunctive Therapy in Patients With Pulmonary Evolution Tuberculosis
Acronym: VitaminD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Martha Torres Rojas, Chairwoman of Microbiology Research Department, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INERC50-13
Record Dates: First submitted 2014-11-12; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The patient will take a single tablet of placebo daily for 60 days. Each patient will go to the hospital in order to take the blood sample.
- VitaminD (Experimental): The patient will take a single tablet of Vitamin D (200 International Units) daily for 60 days. Each patient will go to the hospital in order to take the blood sample.
  Interventions: Dietary Supplement: VitaminD

INTERVENTIONS:
Dietary Supplement: VitaminD — 200 International Units (oral dose) daily of 60 days
  Arms: VitaminD

SUMMARY:
Tuberculosis (TB) is the second largest infectious disease that causes death in the last 4 centuries in all the world. Observational studies found an association between vitaminD and TB, suggesting a potential therapeutic role of vitaminD supplementation in patients with active tuberculosis. The hypothesis is that the administration of vitaminD is associated with changes in the levels of cytokines in patients with tuberculosis treated with first-line drugs. The aim of this study is to evaluate the effect of vitaminD supplementation on the clinical course, the time of negative smears and cultures, and the effect on the immune response in patients with pulmonary tuberculosis (TBP).

DETAILED DESCRIPTION:
We are going to include of 60 patients diagnosed with confirmed TBP with and without diabetes mellitus, by positive smear and culture for Mycobacterium tuberculosis sensitive to first-line drugs (rifampicin, isoniazid, pyrazinamide and ethambutol), which will be grouped as follows: 1) patients who receive vitamin D (VD) (n = 30) and 2) patients who not receive vitamin D (NVD) (n = 30) in addition to drug treatment of tuberculosis drug frontline. Blood samples must be taken each month until the end of treatment.The VD group of participants will receive treatment with a daily dose of Vitamin D 200 International Units (IU) during the first two months of treatment. All Patients who participate must give their written consent.

First, we are going to separate the peripheral blood mononuclear cells with Ficoll reagent. Then, for the determination of intracellular cytokines in basal conditions and after the antigenic stimulation with M.tuberculosis, the flow cytometric technique is going to be used and the results will be analyzing in a flow cytometer. We are going to infected cells with M. tuberculosis strain at a multiplicity of infection (MOI) of 1 and 10, in order to determinate phagocytosis and bactericidal activity of peripheral whole blood of patients, using Colony Forming Units (CFU) and staining. Extraction of RNA will be performed according to the kit supplier. The amplification reaction is going to perform with Applied Biosystems and Sybr Green Master Mix. We are going to use the unpaired Student t test, for the normal distribution parameters.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 and under 65 years old, diagnosed with tuberculosis confirmed by positive smear and positive culture, without documented evidence of previous treatment for TB, with hemoglobin values greater than 10 g / dL, and written concent.

Exclusion Criteria:

* Patients diagnosed with HIV, or who do not give written concent, patients with chronic lung disease, patients with clinical evidence of infectious or chronic inflammatory disease processes such as; rheumatoid arthritis, patients with chronic lung disease, systemic lupus erythematosus (SLE), Sjögren Sx, dermatomyositis, scleroderma, seronegative arthritis, gout, inflammatory bowel disease, chronic active hepatitis, glomerulonephritis, rheumatic fever and patients with cardiac disease, cancer, and patients with a history of alcohol or drug abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Determination of cytokines | 6 months
  First, we are going to separate the peripheral blood mononuclear cells with Ficoll reagent. Cells were adjusted and placed in 1 mL tubes, with an antibody will be incubated for 15 min. at room temperature. Anti-antibody corresponding isotypes are going to incubate for 20 min at room temperature. The cells are going to be fixed with 1% paraformaldehyde before acquiring and analyzing in the flow cytometer. The concentration of Interleucin 17 (IL-17), Interferon-g and Tumor Necrosis Factor-a in culture supernatants of infected cells in vitro with M.tuberculosis are going to be measure. We are going to determinate them by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Edith Escudero, Degree, Study Director — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- Martha Torres Rojas, Mexico City, Mexico City, Mexico

REFERENCES:
- [Result] Gibney KB, MacGregor L, Leder K, Torresi J, Marshall C, Ebeling PR, Biggs BA. Vitamin D deficiency is associated with tuberculosis and latent tuberculosis infection in immigrants from sub-Saharan Africa. Clin Infect Dis. 2008 Feb 1;46(3):443-6. doi: 10.1086/525268. PMID 18173355
- [Result] Nnoaham KE, Clarke A. Low serum vitamin D levels and tuberculosis: a systematic review and meta-analysis. Int J Epidemiol. 2008 Feb;37(1):113-9. doi: 10.1093/ije/dym247. PMID 18245055
- [Result] Martineau AR, Timms PM, Bothamley GH, Hanifa Y, Islam K, Claxton AP, Packe GE, Moore-Gillon JC, Darmalingam M, Davidson RN, Milburn HJ, Baker LV, Barker RD, Woodward NJ, Venton TR, Barnes KE, Mullett CJ, Coussens AK, Rutterford CM, Mein CA, Davies GR, Wilkinson RJ, Nikolayevskyy V, Drobniewski FA, Eldridge SM, Griffiths CJ. High-dose vitamin D(3) during intensive-phase antimicrobial treatment of pulmonary tuberculosis: a double-blind randomised controlled trial. Lancet. 2011 Jan 15;377(9761):242-50. doi: 10.1016/S0140-6736(10)61889-2. Epub 2011 Jan 5. PMID 21215445
- See also: World Health Organization webpage. — http://www.who.int/tb/publications/global_report/en/.